CLINICAL TRIAL: NCT01017159
Title: Randomised, Double-blinded, Placebo-controlled Trial of Subcutaneous Immunoglobulin Treatment in Patients With Chronic Inflammatory Demyelinating Polyradiculoneuropathy (CIDP)
Brief Title: Subcutaneous Immunoglobulin Treatment of Patients With Chronic Inflammatory Demyelinating Polyradiculoneuropathy (CIDP)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of Aarhus (Other)
Collaborators: Baxter Healthcare Corporation (Industry); GCP-unit at Aarhus University Hospital, Aarhus, Denmark (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: EudraCT number: 2009-013930-25
Record Dates: First submitted 2009-11-06; First posted 2009-11-20 (Estimated); Last update posted 2011-11-10 (Estimated); Status verified 2011-11

CONDITIONS: Polyradiculoneuropathy, Chronic Inflammatory Demyelinating
Keywords: Polyradiculoneuropathy, Chronic Inflammatory Demyelinating; Subcutaneous immunoglobulin
MeSH Terms: conditions — Polyradiculoneuropathy, Chronic Inflammatory Demyelinating

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Subcutaneous immunoglobulin (Active Comparator)
  Interventions: Drug: Subcutaneous immunoglobulin
- Saline (Placebo Comparator)
  Interventions: Drug: Subcutaneous immunoglobulin

INTERVENTIONS:
Drug: Subcutaneous immunoglobulin — The subcutaneous immunoglobulin is infused in the subcutaneous tissue on the abdomen twice or thrice a week, with a maximal speed of 2 mL/h. Every time 20 mL is infused, the needle is removed to a new place.
  Other Names: Subcuvia®

SUMMARY:
The purpose of this study is to determine whether subcutaneous immunoglobulin given in small doses, is effective in maintaining the force, in patients with chronic inflammatory demyelinating polyradiculoneuropathy compared with placebo (saline infusions), and intravenous immunoglobulin.

DETAILED DESCRIPTION:
CIDP is an autoimmune disease of the peripheral nervous system, responding well to treatment with intravenous immunoglobulin (IVIg), steroids and plasmapheresis. IVIg is effective in treating patients with CIDP, but most of the patients need long time maintenance treatment, which is associated with decreased autonomy and regular hospital admissions. Furthermore many of the patients complain of infusion related side effects such as headache, chills and fatigue, and over time there is problems obtaining intravenous entry because of occlusion of the veins.

There is therefore a critical need for alternative methods to IVIg treatment. The aim of this study is to evaluate the efficacy, tolerability and safety of small doses of immunoglobulin administered subcutaneously (SCIg), compared with placebo. At the same time we compare the efficacy of SCIg with the regular IVIg treatment.

We therefore hypothesize, 1: SCIg is better than subcutaneous placebo infusions, and is as good as IVIg in maintaining muscle function in patients with CIDP. 2: SCIg home treatment is safe and tolerable. 3: SCIg home treatment is preferred to IVIg under hospital admission, by the patients.

ELIGIBILITY:
Inclusion Criteria:

* All patients with typical or pure motor CIDP, who meet the clinical or electrophysiological criteria of the EFNS/PNS for certain or probable CIDP and who are in regular treatment with IVIg on one of the neurological departments in Denmark, are eligible for the study

Exclusion Criteria:

* Pregnancy
* Known cancer disease
* Severe medical diseases
* Other immuno modulating treatment than low-dose steroid (prednisolone < 25 mg/day) within the last 6 weeks before inclusion
* Hepatitis B or C or HIV
* Breast-feeding
* Non-responding to treatment with intravenous immunoglobulin
* Known hypersensitivity to intravenous immunoglobulins or Kiovig

Adverse events:

* Previous moderate headache or minor rash for a few days during or after infusion is not an exclusion criteria
* In case of severe adverse effects to treatment patients are excluded. Moderate or mild side-effects can be treated with analgetics or steroids for 1-2 weeks during the initial study phase

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2010-04; Primary Completion 2011-11 (Actual); Study Completion 2011-11 (Actual)

PRIMARY OUTCOMES:
Strength assessed by isokinetic strength measurements, in the active treatment group compared with the placebo group. | The study period is 98 days. Isokinetic strength will be measured on day 14, 28, 84 and 98 of the study period. If there is a drop-out before day 84, the strength measurement will take place on this day, and the last two measurements will be left out.

SECONDARY OUTCOMES:
Efficacy and feasibility of subcutaneous immunoglobulin infusions. | Feasibility will be recorded continously in a patient diary and in the CRF (case report form), and efficacy will be calculated at the end of the study, after approximately three months.

CONTACTS AND LOCATIONS:
Overall Officials: Johannes Jakobsen, Dr., MD, Principal Investigator
Locations (1):
- Aarhus University Hospital, Noerrebrogade, Department of Neurology, Aarhus, Aarhus, Denmark